CLINICAL TRIAL: NCT07197970
Title: A Prospective, Multi-center, Randomized Controlled, Clinical Trial to Evaluate the Safety and Efficacy of NxiDIME™ Intracranial Drug-eluting Self-expanding Stent System
Brief Title: Drug- Eluting Stent for Symptomatic Intracranial Arterial Stenosis
Acronym: DESIAS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Feng Gao, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QX2025-002-01
Record Dates: First submitted 2025-09-25; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-04

CONDITIONS: Symptomatic Intracranial Atherosclerotic Stenosis
Keywords: symptomatic intracranial atherosclerotic stenosis; Drug-Eluting Stent; strok

STUDY DESIGN:
Intervention Model Description: This investigation is a prospective, multicenter, randomized controlled, non-inferiority clinical trial, to evaluate the safety and efficacy of the NxiDIME™ Intracranial drug-eluting self-expanding stent against the NOVA DES® Intracranial Drug-Eluting balloon-expandable stents for patients with symptomatic intracranial atherosclerotic stenosis.
Masking Description: Prospective randomized open blinded end-point (PROBE) study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Endovascular angioplasty with NxiDIME™ Intracranial Drug-Eluting self-expanding Stent System
  Interventions: Device: NxiDIME™ Intracranial Drug-Eluting Stent System
- Controal group (Active Comparator): Endovascular angioplasty with NOVA Intracranial Drug-Eluting Balloon-expandable Stent
  Interventions: Device: NOVA DES Intracranial Drug-Eluting Stent

INTERVENTIONS:
Device: NxiDIME™ Intracranial Drug-Eluting Stent System — The experimental group will receive the NxiDIME™ Intracranial Drug-Eluting self-expanding Stent System (RICOTON Technology Co., Ltd.)
  Arms: Experimental group
Device: NOVA DES Intracranial Drug-Eluting Stent — The experimental group will receive the NOVA DES Intracranial Drug-Eluting balloon-expandable stent System
  Arms: Controal group

SUMMARY:
This investigation is a prospective, multicenter, randomized controlled, non-inferiority clinical trial, to evaluate the safety and efficacy of the investigational device against alternative models/specifications of the control device. The study will be conducted across multiple Chinese centers, with planned enrollment of 224 patients with symptomatic intracranial atherosclerotic stenosis. Subjects meeting all inclusion criteria and without any exclusion criteria will enter the investigation after providing written informed consent via ethics committee-approved informed consent forms (ICFs). The randomized controlled study plans to enroll 224 patients, stratified by intracranial lesion location (anterior/posterior circulation), through a centralized randomization system. The experimental group will receive the NxiDIME™ Intracranial Drug-Eluting Stent System (RICOTON Technology Co., Ltd.), while the control group will receive the NOVADES® Intracranial Drug-Eluting Stent System.

All subjects underwent follow-up visits on the day of the procedure, within 7 days postoperatively or prior to discharge, and at 30 days, 6 months, and 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and ≤ 80 years old, regardless of gender.
2. Symptomatic intracranial arterial stenosis (TIA/ischemic stroke within 180 days attributed to intracranial arteries including the intracranial internal carotid artery, middle cerebral artery, intracranial vertebral artery, or basilar artery, with stenosis severity ≥70% and ≤99% measured by DSA using WASID criteria), currently receiving at least one antiplatelet therapy;
3. Poor collateral circulation or hypoperfusion in the target vessel territory (Poor collateral circulation: American Society of Interventional and Therapeutic Neuroradiology/Society of Interventional Radiology (ASITN/SIR) score < 3; Hypoperfusion: 1. The cerebral blood flow (CBF) in the target artery territory decreases by > 30% during CT or magnetic resonance perfusion imaging (MR perfusion); or 2. There are hemodynamic ischemic lesions on MRI or CT, such as watershed infarction);
4. Target lesion vessel diameter 1.0-5.5 mm with lesion length ≤40 mm (If: 2.25 mm ≤ target vessel diameter ≤4.0 mm and lesion length ≤15 mm, enroll in randomized controlled study; 1.0 mm ≤ target vessel diameter <2.25 mm or 4.0 mm < target vessel diameter ≤5.5 mm or 15 mm < lesion length ≤40 mm, enroll in single-arm cohort study);
5. mRS score ≤ 2;
6. Patient or legal guardian voluntarily participates and signs the written ICF, with willingness to comply with protocol-specified examinations and follow-up.

Exclusion Criteria:

1. History of prior stent implantation or surgical treatment at the target lesion;
2. Intracranial hemorrhage within 30 days preoperatively or presence of untreated chronic subdural hematoma ≥5 mm;
3. Major surgical procedure within 30 days prior to the procedure;
4. Acute ischemic stroke within 14 days prior to the procedure;
5. Symptomatic carotid stenosis ≥50% outside the target lesion, or coexisting intracranial/extracranial vascular stenosis ≥70% requiring intervention;
6. Severe calcification, significant stenosis, or tortuosity of the target vessel precluding device deployment as assessed by investigators;
7. Intracranial tumor, arteriovenous malformation, or tandem aneurysms proximal/distal to the target lesion;
8. Non-atherosclerotic stenosis etiology (e.g., arterial dissection, moyamoya disease, vasculitis);
9. Cardiac thromboembolic sources (e.g., atrial fibrillation, left ventricular thrombus, myocardial infarction within 6 weeks);
10. Uncontrolled hypertension (persistent systolic blood pressure (SBP) ≥180 mmHg or diastolic blood pressure (DBP) ≥110 mmHg);
11. Contraindications to antiplatelet/anticoagulant therapy, coagulopathy or bleeding diathesis precluding intervention per investigator judgment;
12. Severe comorbidities: cardiac failure (New York Heart Association (NYHA) Class III-IV), respiratory/renal failure (serum creatinine >3.0 mg/dL (264 μmol/L)), Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) more than 3 times the upper limit of the normal value), active malignancy;
13. Hypersensitivity to rapamycin, polylactic-co-glycolic acid, nitinol, platinum-tungsten, anesthetics, or contrast agents;
14. Life expectancy <1 year;
15. Pregnancy, lactation, or planned pregnancy within 1 year;
16. Concurrent participation in other clinical trials without completing primary endpoint follow-up;
17. Cognitive impairment or psychiatric disorders compromising protocol compliance; other exclusionary conditions per investigator discretion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
12-month incidence rate of in-stent restenosis | 12-month
  In-stent restenosis is defined as luminal stenosis >50% within the stent or adjacent 5-mm segments, accompanied by late lumen loss >20% relative to immediate post-procedural measurements by follow-up DSA.

CONTACTS AND LOCATIONS:
Locations (1):
- A prospective, multi-center, randomized controlled, non-inferiority clinical trial to evaluate the safety and efficacy of the NxiDIME™ Intracranial Drug-Eluting Stent System in the treatment of symptomatic intracranial atherosclerotic stenosis lesions, Beijing, Beijing Municipality, China